CLINICAL TRIAL: NCT05167136
Title: "Green Hospital" Awareness Level and Satisfaction of Health Practitioners - A Private Hospital Experience in Turkey
Brief Title: Green Hospital Awareness
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: ILKE KUPELI (Other)
Responsible Party: Sponsor-Investigator, ILKE KUPELI, investigator, Biruni University
Organization: Biruni University (Other)
Other Study IDs: BIRUNI 3
Record Dates: First submitted 2021-11-18; First posted 2021-12-22 (Actual); Last update posted 2021-12-22 (Actual); Status verified 2021-12

CONDITIONS: Satisfaction, Personal
MeSH Terms: conditions — Personal Satisfaction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Awareness Level — Demands and expectations about the green hospital were measured with a questionnaire applied to 287 people, consisting of health professionals and employees in a small private hospital that does not have a "green hospital" certificate in the province of Istanbul.

SUMMARY:
Environmentally conscious hospitals plan their designs as green hospitals and aim to use resources efficiently. Green buildings are defined as buildings that respect nature, are ecological, comfortable and reduce energy consumption. The aim of our study is to investigate the awareness level and satisfaction of the employees of a small private hospital in the city center without a "green hospital" certificate regarding the "green hospital" elements.

ELIGIBILITY:
Inclusion Criteria:

* consisting of health professionals and employees
* working in a small private hospital that does not have a "green hospital" certificate

Exclusion Criteria:

* who refused to participate in the survey

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 280 people, consisting of health professionals and employees in a small private hospital that does not have a "green hospital" certificate in the province of Istanbul.
Sampling Method: Non-Probability Sample
Enrollment: 280 (Estimated)
Dates: Start 2021-12-18 (Estimated); Primary Completion 2021-12-30 (Estimated); Study Completion 2022-01-15 (Estimated)

PRIMARY OUTCOMES:
level of awareness | 15 DAYS
  A 5-point Likert type scal

CONTACTS AND LOCATIONS:
Locations (1):
- Ilke Kupeli, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Abbaszadeh, S., Zagreus, L., Lehrer, D., Huizenga, C. (2006). Occupant Satisfaction with Indoor Environmental Quality in Green Buildings. Proceedings of Healthy Buildings. 3: 365-370.
- [Result] Khairunnisa, R. A., Ulfa, M., Azizi, M. R., & Setyonugroho, W. (2021). A FUTURE GREEN AND HEALTHY HOSPITAL: A REVIEW ARTICLE. Proceedings of International on Healthcare Facilities, 1(1), 82-94